CLINICAL TRIAL: NCT06508541
Title: The Prognosis of Colorectal Cancer Patients After Indocyanine Green Fluorescence-guided Radical Surgery: a Retrospective Cohort Study
Brief Title: The Prognosis of Colorectal Cancer Patients After Indocyanine Green Fluorescence-guided Radical Surgery
Status: Completed | Type: Observational
Sponsor: Shanghai Tong Ren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-06-001
Record Dates: First submitted 2024-07-13; First posted 2024-07-18 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer
Keywords: Indocyanine green; Colorectal cancer; prognosis
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Routine surgical specimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- conventional surgery: All patients underwent standard complete mesocolic excision (CME) or total mesorectal excision (TME) with curable purpose.
  Interventions: Procedure: conventional surgery
- Indocyanine green fluorescence-guided surgery: Approximately 0.3 ml of ICG dissolved in 2.5 mg/ml of sterile water was injected submucosally by the endoscopic doctors through colonoscopy at two points around the tumor.All patients underwent standard complete mesocolic excision (CME) or total mesorectal excision (TME) with curable purpose using ICG lymphangiography procedure
  Interventions: Procedure: ICG Guided surgery; Procedure: conventional surgery

INTERVENTIONS:
Procedure: ICG Guided surgery — In ICG guided surgery group,Approximately 0.3 ml of ICG dissolved in 2.5 mg/ml of sterile water was injected submucosally by the endoscopic doctors through colonoscopy at two points around the tumor.All patients underwent standard complete mesocolic excision (CME) or total mesorectal excision (TME) with curable purpose using ICG lymphangiography procedure
  Groups: Indocyanine green fluorescence-guided surgery
Procedure: conventional surgery — All patients underwent standard complete mesocolic excision (CME) or total mesorectal excision (TME) with curable purpose

SUMMARY:
Previous studies of Indocyanine green (ICG) in colorectal surgery have focused on lymphatic mapping, lymph node detection, and the number of harvested lymph nodes. However, relatively few studies have evaluated the outcomes of this imaging technology, especially the prognosis following of colorectal cancer resection. The present study assessed the prognosis of colorectal cancer patients following ICG fluorescence-guided surgery as compared to conventional surgery without the use of ICG Fluorescence imaging

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years,
* confirmed diagnosis of primary CRC,
* preoperative tumor stage of cT1 to cT4, N-/+, M0 as determined by contrast-enhanced computed tomography (CT),
* no distant metastasis, -American Society of Anesthesiologists(ASA)Physical Status Classification score of 1, 2, or 3-

Exclusion Criteria:

* history of previous colorectal surgery, emergent surgery, or palliative resection;
* pregnancy or breastfeeding;
* allergy or history of an adverse reaction to ICG; and
* severe mental disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with newly diagnosed CRC who underwent CRC surgery between December 2016 and August 2021 in Shanghai Tongren hospital
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
disease-free survival(DFS) | 1 month
  the duration from radical surgery to the confirmation of recurrence or metastasis by regular or telephone follow-up

SECONDARY OUTCOMES:
the number of harvested lymph nodes | 1month
  the number of harvested lymph nodes including positive and negative ones

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tongren Hospital, Changning, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided